CLINICAL TRIAL: NCT02471495
Title: A Multicenter, Single-Arm Study Evaluating the Efficacy of Synergo® Radiofrequency-Induced Thermochemotherapy Effect With Mitomycin C in Non-Muscle Invasive Bladder Cancer Patients With BCG-refractory CIS
Brief Title: RITE-EUROPE (Radiofrequency-Induced Thermochemotherapy Effect-EUROPE)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Enterprises Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RITE-2
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Bladder Cancer
Keywords: NMIBC; Non-Muscle-Invasive Bladder Cancer; Nonmuscle Invasive Bladder Cancer; BCG refractory; BCG failure; Carcinoma in situ; CIS
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Carcinoma in Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Synergo® RITE + MMC (Experimental): Induction
  Patients will receive 8 weekly treatments of Synergo® RITE + MMC, using the Synergo® System. Each treatment lasts about 60 minutes and consists of two 30-minute cycles with 40 mg MMC/50 ml sterile water for injection each cycle. These 8 treatments will be followed by a pause (see Table 1), after which a follow-up cystoscopy (first follow-up control) will be conducted during Weeks 12-13 (from the first treatment).
  Maintenance
  Patients will receive one Synergo® RITE + MMC treatment every 6 weeks. Each treatment lasts about 60 minutes and consists of two 30-minute cycles with 40 mg MMC/50 ml sterile water for injection each cycle. Maintenance treatments will be given until the end of 12 months after the patient's first induction treatment.
  Interventions: Device: Synergo® RITE + MMC

INTERVENTIONS:
Device: Synergo® RITE + MMC — Synergo® system delivers homogenous microwave hyperthermia to the bladder wall in combination with bladder instillation of cold chemotherapeutic agent - Mitomycin C (MMC).The energy-delivering unit and the intravesical irrigation system are computer-controlled, The irrigation system consists of a disposable tubing line and catheter set. The catheter is a triple-lumen, silicone, transurethral Foley-type catheter.
  MMC is constituted as a powder (40 mg) dissolved in 50 ml sterile water for injection.

SUMMARY:
This multicenter, prospective, single-arm, phase 3 study will assess the proportion of disease-free patients, starting from administration of the first study treatment to at least 12-months after the first treatment, and up to 2 years (the latter only in patients choosing to participate in longer-term disease-free-survival data collection).

DETAILED DESCRIPTION:
The study will consist of three periods: 1) Screening; 2) Induction, and 3) Maintenance treatment and follow-up.

Screening period After signing informed consent, patients will be screened for study eligibility by assessment of inclusion and exclusion criteria. Screening procedures will include collection of demographic data, medical history, physical examination, vital signs, and laboratory evaluations.

Induction period Patients will receive 8 weekly treatments of RITE + MMC, using the Synergo® System. Each treatment lasts about 60 minutes and consists of two 30-minute cycles with 40 mg MMC/50 ml sterile water for injection each cycle. These 8 treatments will be followed by a pause (see Table 1), after which a follow-up cystoscopy (first follow-up control) will be conducted during Weeks 12-13 (from the first treatment).

Maintenance Treatment and Follow-up Period

During the maintenance period, patients will receive one Synergo® RITE + MMC treatment every 6 weeks. Each treatment lasts about 60 minutes and consists of two 30-minute cycles with 40 mg MMC/50 ml sterile water for injection each cycle. Maintenance treatments will be given until the end of 12 months after the patient's first induction treatment, unless the patient's participation in the study is terminated due to either:

1. a lack of complete response (at 6 months) or worsening of disease (at 3 months; see first and second follow-up control below), or
2. recurrence/progression Patients will be assessed by cystoscopy, urine cytology and, if required, subsequent biopsy or transurethral resection (TUR) of suspect areas every 3 months till the end of the study.

Two consecutive definite positive urine cytologies will be required to confirm persistent or recurrent disease if visual and biopsy are negative. In such cases, investigation of extravesical locations (CT-IVU, prostatic urethra biopsy) will be performed between the first and second urine cytology.

At the first follow-up control, i.e., 3 months after administration of the first study treatment, patients will undergo a cystoscopy evaluation.

Patients failing to achieve a disease-free state at the time of the first follow-up will continue in the study, unless a new occurrence of a T1 and/or high-grade lesion is found or any extra-bladder involvement is evident from pathological analysis.

At the second, i.e., 6-month, follow-up visit, patients will undergo biopsies of suspicious areas and random bladder biopsies of the trigone, bladder dome, right, left, anterior and posterior of the bladder wall. Upper tract washes will be performed in patients in whom urine cytology will be positive with no pathological evidence of NMIBC lesions in the bladder or the prostatic urethra. Patients failing to achieve a disease-free state at the time of the 6 month assessment and/or experiencing a new disease occurrence, demonstrated by cystoscopy and biopsy, and/or in whom extra-bladder involvement is suggested by a positive upper tract washes result will be removed from the study.

Upper tract imaging (CT-IVU imaging is recommended, IVU if CT not available) will be performed at 12 months from the first study treatment.

Extended treatment and follow-up period For longer-term disease-free-survival data collection purposes, patients free of tumor at the end of the study will be offered to continue receiving one Synergo® RITE + MMC treatment every 8 weeks. Each such treatment will last about 60 minutes and will consist of two 30-minute cycles with 40 mg MMC/50 ml sterile water for injection, each cycle. These treatments will be given until the end of 24 months after the patient's first induction treatment. See table 2 for details on the extended treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CIS, with or without coexisting papillary NMIBC, who either:

   * fail to achieve a disease-free status by 6 months after initial BCG therapy, with maintenance or re-induction at 3 months due to either persistent or rapidly recurrent disease, or
   * experience a worsening in NMIBC state following initial BCG therapy presenting with a new NMIBC instance, other than TaLG.
2. All clinical, intra-operative and pathological items for the EAU risk stratification must be documented including a bladder map.
3. Patients with papillary disease must have undergone a repeat TUR:

   * if the initial TUR was incomplete.
   * if there was no muscle in the specimen after the initial TUR (except in TaLG tumors).
   * in all T1 tumors. TUR of T1 sites must include muscle.
   * in all HG tumors > 3cm.
4. CT-IVU or IVU confirmation of absence of tumor(s) in the upper tract, kidney and ureters performed within 6 months before the treatment initiation in selected cases as recommended in latest EAU guidelines published prior to screening. If IVU protocol not available or contrast allergy/poor renal function preclude such imaging, then non-contrast CT or MRI of the abdomen/pelvis within the same timeframe will suffice.
5. Visual inspection to exclude urothelial carcinoma (UC) in the urethra during cystoscopy.
6. Biopsy of the prostatic urethra in male patients prior to recruitment to exclude UC of the prostatic urethra, in patients with:

   * tumor of trigone,
   * tumor of bladder neck, or
   * abnormal prostatic urethra
7. All patients must have urine cytology collected from either voided urine or bladder wash within the screening period prior to recruitment.
8. All patients must have prostatic urethral biopsies collected within the screening period prior to recruitment.
9. Age ≥ 18 yrs.
10. Normal kidneys and ureters.
11. Pre-treatment hematology and biochemistry values within the limits:

    * Hemoglobin ≥ 10 g/dl
    * Platelets ≥ 150 x 10^9/L
    * WBC ≥ 3.0 x 10^9/L
    * ANC ≥ 1.5 x 10^9/L
    * Serum creatinine < 1.5 x ULN
    * SGOT < 1.5 x ULN
    * SGPT < 1.5 x ULN
    * Alkaline phosphatase < 1.5 x ULN
12. Negative pregnancy test for women of childbearing potential.
13. A life expectancy at least of the duration of the study (up to 13 months).
14. Patients unfit or unwilling to have a full or partial (if appropriate) cystectomy.
15. Signed informed consent.

Exclusion Criteria:

1. Non-UC tumor of the urinary tract.
2. Upper tract and intramural tumors (e.g., in ostium).
3. Positive selective cytology from the upper tract.
4. History of stage > T1 UC.
5. Papillary tumor in repeat TUR in patients diagnosed with HG > 3cm and/or T1 in the initial TUR.
6. Papillary tumor ≥ T1 in repeat TUR
7. Known or suspected reduced bladder capacity. Patients will have a US estimation of maximum bladder capacity or void spontaneously the maximum they can retain in their bladder, and this will be used to determine urine volume. A minimum volume of 250 ml is required.
8. Bleeding disorder.
9. Macrohematuria of ≥ 250 RBC/uL or equivalent (e.g., > "+++" erythrocytes in a dipstick analysis) within 4 weeks before treatment start.
10. Lactating women.
11. Women of childbearing potential unwilling or unable to use adequate contraception if sexually active.
12. More than a maintenance dose of oral corticosteroids (maintenance dose is defined as the same dose regimen over the past 6 months for a condition requiring continual corticosteroid treatment) or patients with an immunocompromised state for any reason.
13. More than low-dose methotrexate (>17.5 mg once a week).
14. Other malignancy within the past 5 years, except: non-melanomatous skin cancer cured by excision, surgically treated carcinoma in situ of the cervix or ductal CIS (DCIS)/lobular CIS (LCIS) of the breast or stable prostate cancer (under active surveillance or hormone control) with a life expectancy of more than 5 years.
15. Any known allergy (e.g., to MMC) or adverse event that would prevent a prospective study participant from receiving the study treatment.
16. Known untreated urethral strictural disease or bladder neck contracture or any other condition that may prevent catheterization with 21F catheter. Patients may undergo dilation or urethral incision before entering the study.
17. Bladder diverticula with cumulative diameter > 1cm or tumor in a diverticulum.
18. UTI at any time within 4 weeks before treatment start.
19. Significant urinary incontinence (spontaneous, requiring use of pads).
20. History of pelvic irradiation.
21. Patients with implanted electronic devices (such as cardiac pacemakers) unless they receive permission from their treating physician (e.g., cardiologist) and are monitored by a treating physician during the treatment session.
22. Participation in another study, unless discussed with and approved by the study manager.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 12 months
  The study will be deemed successful if the recurrence-free survival probability after 12 months is at least 30%.

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | 6 months after first treatment
  A satisfactory outcome will be if the CRR at 6 months is at least 40%.
Rate of serious adverse events | 12 months
Proportion of patients who discontinue treatment for safety reasons. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Igal Ruvinsky, PhD, Study Director — Medical Enterprises; Shariat Shahrokh, Prof. med, Principal Investigator — Medical University Vienna, General Hospital

IPD SHARING:
Plan to Share IPD: No